CLINICAL TRIAL: NCT05139342
Title: Evaluation of the Efficacy of a Two-week Expiratory Muscle Training on Swallowing Function in Patients With Parkinsonian Disorders
Brief Title: Evaluation of the Efficacy of a Two-week EMST on Dysphagia in Parkinsonian Patients
Acronym: EMST-PS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kliniken Beelitz GmbH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-2155-BO-ff
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Parkinson Disease; Multiple System Atrophy; Progressive Supranuclear Palsy
Keywords: Parkinson's disease; Multiple System Atrophy; 4repeat tauopathies; dysphagia; EMST; FEES
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD patients (Active Comparator): patients diagnosed with PD will be allocated to this arm
  Interventions: Device: expiratory muscle strentgh training (EMST)
- MSA patients (Active Comparator): patients diagnosed with MSAwill be allocated to this arm
  Interventions: Device: expiratory muscle strentgh training (EMST)
- 4RT patients (Active Comparator): patients diagnosed with 4RT will be allocated to this arm
  Interventions: Device: expiratory muscle strentgh training (EMST)

INTERVENTIONS:
Device: expiratory muscle strentgh training (EMST) — All patients undergo EMST training, and results will be compared between groups.
  After individual adjustment of the EMST device for each patient, the patient receives speeach adn instruction from a speech and language pathologist on the correct use of the EMST device. The intervention regime then consists of 5x5 breaths per day for 14 consecutive days.

SUMMARY:
This is an interventional therapy study designed to evaluate the efficacy of a two-week intervention, i.e. training with a specialized exhalation training device (called expiratory muscle strength training; EMST150 or EMST75; Aspire Products, Gainsville, FL) on swallowing function in patients with neurodegenerative Parkinsonian disorders. This study involves a routine endoscopic evaluation of swallowing (FEES) to diagnose dysphagia before and after the intervention. Between the two FEES, a two-week exhalation training program takes place, which the patients perform independently following instructions from a speech and lanuage pathologist. In addition demographic and disease-specific data and two questionnaires (Swallowing Disturbance Questionnaire for Parkinson's disease patients, SDQ-PD, and Swallowing specific Quality Of Life Questionnaire SWAL-QoL) are recorded.

DETAILED DESCRIPTION:
This is an interventional therapy study designed to evaluate the efficacy of a two-week intervention, i.e. training with a specialized exhalation training device (called expiratory muscle strength training; EMST150 or EMST75; Aspire Products, Gainsville, FL) on swallowing function in patients with neurodegenerative Parkinsonian disorders. This study involves a routine endoscopic evaluation of swallowing (FEES) to diagnose dysphagia before and after the intervention. Between the two FEES, a two-week exhalation training program takes place, which the patients perform independently following instructions from a speech and lanuage pathologist. In addition demographic and disease-specific data and two questionnaires (Swallowing Disturbance Questionnaire for Parkinson's disease patients, SDQ-PD, and Swallowing specific Quality Of Life Questionnaire SWAL-QoL) are recorded.

Main hypothesis: Two weeks of EMST will lead to a significant improvement of the endoscopic dysphagia score in patients with neurodegenerative Parkinsonian disorders with endoscopically proven oropharyngeal dysphagia. Patients with idiopathic Parkinson's syndrome as well as its differential diagnoses, multiple system atrophy (MSA) and diseases from the group of 4repeat tauopathies, will be examined.

Idiopathic Parkinson's disease (PD):

More than 80% of all patients with PD develop clinically relevant dysphagia during the course of the disease. This can lead to a significant reduction in quality of life, decreased medication efficacy, malnutrition, dehydration, and ultimately aspiration pneumonia in affected patients, which is the most common cause of death in advanced PD patients. The cause of PD-associated dysphagia is a multifactorial genesis with impairment of dopaminergic and non-dopaminergic pathways of the central swallowing network and additional peripheral neuromuscular influences.

Multiple System Atrophy (MSA):

MSA is clinically associated with autonomic dysregulation manifested by neurogenic urinary bladder emptying dysfunction, orthostatic hypotension, sleep-related respiratory dysregulation, etc. in addition to Parkinsonian and/or cerebellar symptoms. Median survival after diagnosis is approximately 7 years. At disease onset, differentiation from idiopathic PD is difficult. However, relatively early in the course of the disease, symptoms such as a brittle voice or stridor may appear during normal breathing, which may be clues to the diagnosis of MSA. Since laryngeal abnormalities are associated with a significantly reduced life expectancy, they require special attention and diagnosis. In this regard, we have recently shown that a high prevalence of laryngeal movement abnormalities is present in MSA patients and can even be used to differentiate them from idiopathic Parkinson's disease. Swallowing function, the regulation of which is associated with autonomic centers of laryngeal function, is also often impaired early in patients with MSA. Because dysphagia can further limit quality of life and life expectancy, this symptom also requires early diagnosis and treatment. We could recently show that the dysphagia pattern also differs between PD and MSA.

4repeat tauopathies (4RT): The form of 4RT, also named progressive supranuclear gaze palsy (PSP) with all clinical subtypes, is a rapidly progressive neurodegenerative disease that leads to progressive functional impairment of cortical and subcortical function in affected individuals due to accumulation of tau protein in the brain. Due to the clinical variability of presentation, early diagnostic certainty is desirable, especially since human IgG4- antibodies directed against extracellular tau protein are currently in clinical trials to modify the course of the disease (see NCT03068468, NCT02985879). 4RT are also associated with swallowing and speech problems, and aspiration pneumonia is among the leading causes of death in this disease group. In addition, characteristic abnormalities may also occur due to dystonic dysinnervation of laryngeal muscles.

For dysphagia in atypical Parkinsonian syndromes, there are no proven interventional or drug therapy options. Previous studies in patients with PD had shown efficacy of a four-week training with a special expiratory muscle strength training (EMST) device. Both swallowing reliability and swallowing efficiency were improved. Studies on the efficacy of EMST on dysphagia of atypical Parkinsonian syndromes do not yet exist. Having demonstrated the efficacy of EMST in a 4-week intervention regime, the first aim is to test whether a shortened intervention duration of two weeks is also effective in patient with PD. In addition, this protocol will be performed in patients with MSA and 4RT to investigate effects, particularly on swallowing safety (reduction of penetration/aspiration events) and swallowing efficiency (reduction of pharyngeal residuals). Currently, all patients with PD, MSA, or 4RT at participating study sites receive a speech and language pathology examination and endoscopic diagnostics according to a defined protocol. In addition to phoniatric and swallowing-specific examinations, an endoscopic evaluation of swallowing (FEES) is routinely performed. Regarding the efficacy of EMST training on pharyngeal dysphagia in patients with PD, two randomized, placebo-controlled studies from recent years with n=60 and n=50 patients, respectively, have already shown an efficacy of training on both swallowing reliability and swallowing efficiency in PD patients. Relevant side effects or risks from training for the patients were not reported in the studies.

Studies using an EMST device have been conducted in recent years not only in patients with IPS, but also in patients with dysphagia due to other primary pathologies (e.g., amyotrophic lateral sclerosis, multiple sclerosis, stroke, etc.). In summary, a positive effect was shown, particularly on laryngeal muscle strengthening, which was reflected in an improvement in dysphagia.

The affected patients receive an initial endoscopic evaluation of the swallowing act in the clinical setting as part of routine diagnostics. In addition, oral and written patient education is provided. After written consent on the informed consent form, the following data are then collected anonymously prior to the start of the intervention:

1. sociographic data
2. disease milestones
3. MDS-UPDRS I-IV
4. UMSARS / PSP-RS
5. SDQ-PD
6. SWAL-QOL
7. Hoehn and Yahr stage
8. Current drug therapy
9. MSA-FEES examination protocol
10. Pulmonary function test

This is followed by the individual adjustment of the EMST device for the respective patient. For this purpose, the maximum expiratory pressure (MEP) is first determined for the respective patient in the pulmonary function examination using a pressure manometer. 75% of the MEP is set for the subsequent training on the EMST device. This is then followed by the actual intervention. For this, the patient receives logopedic instruction on the correct use of the EMST device. The intervention regime then consists of 5x5 breaths per day for 14 consecutive days. Immediately following, items 3-10 will be collected again.

1. The collection of data regarding the effectiveness of EMST in a shortened protocol (two weeks) on swallowing function in patients with PD can help to integrate this form of therapy firmly in the therapy regime of speech and language therapy also in the context of inpatient stays.
2. The evaluation of the efficacy of EMST in atypical Parkinsonian syndromes is the first interventional study with the attempt to improve dysphagia in these disease spectra. If this study demonstrates improvement in dysphagia in MSA and 4RT, appropriate patients would be offered a specific EMST in the future, which may then delay or prevent the development of higher-grade dysphagia. Since consecutive aspiration pneumonia on the floor of neurogenic dysphagia is the leading cause of death in these patients, this could at least delay serious medical complications in the future, improve quality of life, and prolong survival. In addition, new evidence would be gained for the use of activating therapies in the treatment of Parkinson's-associated dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age with.
* diagnosis of idiopathic Parkinson's disease according to the updated diagnostic criteria (Postuma 2015) or (3) Diagnosis of a possible or probable Multiple System Atrophy according to the diagnostic criteria (Gilman 2008) or (4) Diagnosis of a possible or probable progressive supranuclear gaze palsy according to the diagnostic criteria (Höglinger 2017) (5) in Hoehn and Yahr stages I-V.

Exclusion Criteria:

1. Patients that do not sign the informed consent form
2. Patients who have contraindications for a fiberendoscopic swallowing examination
3. Patients who have contraindications to the two weeks of EMST training (e.g., severe pulmonary disease, severe dementia).
4. Patients who have competing causes of dysphagia (e.g., history of stroke, tumor in the neck).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
dysphagia-score | 14 days
  improvement of dysphagia score observed on FEES after the intervention in all three groups.
  Three salient parameters of swallowing function are evaluated:
  1. premature spillage
  2. penetration-aspiration events
  3. residue
  The scoring of these parameters is done separately using 3 ordinal 5-point scales (0- 4, from 0 = best to 4 = worst).
  Dysphagia severity, assessed by FEES, is classified according to a four-point scale (0-3) developed for patients with PD and atypical parkinsonism:
  0 = no relevant dysphagia,
  1. = mild dysphagia (premature spillage and/or residues without penetration/aspiration events),
  2. = moderate dysphagia (penetration/aspiration events of one consistency), and
  3. = severe dysphagia (penetration/aspiration events of two or more consistencies).

SECONDARY OUTCOMES:
SDQ-PD score | 14 days
  improvement of SDQ-PD score after the intervention. SDQ comprises 15 items (score range 0.5 - 44.5 with higher scores indicating more severe swallowing disturbance) that are scored either 0 = symptom never appears,
  1. = appears seldom (≤1/month),
  2. = appears often (1-7/week),
  3. = appears very often (>7/week), item 15 was scored dichotomously: yes = 0.5
SWAL-QoL score | 14 days
  improvement of SWAL_QoL score after the intervention
  A 44item questionnaire (range 44 - 220) with lower scores indicating more severe impairment of swallowing-associated quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Florin Gandor, MD, Principal Investigator — Movement Disorders Hospital Beelitz-Heilstätten,
Locations (3):
- Germany (3):
  - Movement Disorders Hospital - Kliniken Beelitz, Beelitz-Heilstätten, Brandenburg
  - Universitätsklinium Münster, Münster
  - Klinikum Osnabrück, Osnabrück

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis, informed consent form, and study data, including de-identified participant data, will be made available to others with publication upon formal request and receipt of a signed material transfer agreement. Requests should be directed to the corresponding author. Data will only be shared via individual secured network connections.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after completion of data collection
Access Criteria: Requests should be directed to the PI. Data will only be shared via individual secured network connections.

REFERENCES:
- [Background] Claus I, Muhle P, Czechowski J, Ahring S, Labeit B, Suntrup-Krueger S, Wiendl H, Dziewas R, Warnecke T. Expiratory Muscle Strength Training for Therapy of Pharyngeal Dysphagia in Parkinson's Disease. Mov Disord. 2021 Aug;36(8):1815-1824. doi: 10.1002/mds.28552. Epub 2021 Mar 2. PMID 33650729
- [Background] Vogel A, Claus I, Ahring S, Gruber D, Haghikia A, Frank U, Dziewas R, Ebersbach G, Gandor F, Warnecke T. Endoscopic Characteristics of Dysphagia in Multiple System Atrophy Compared to Parkinson's Disease. Mov Disord. 2022 Mar;37(3):535-544. doi: 10.1002/mds.28854. Epub 2021 Nov 13. PMID 34773420
- [Background] Brooks M, McLaughlin E, Shields N. Expiratory muscle strength training improves swallowing and respiratory outcomes in people with dysphagia: A systematic review. Int J Speech Lang Pathol. 2019 Feb;21(1):89-100. doi: 10.1080/17549507.2017.1387285. Epub 2017 Nov 1. PMID 29090601
- [Background] Gandor F, Vogel A, Claus I, Ahring S, Gruber D, Heinze HJ, Dziewas R, Ebersbach G, Warnecke T. Laryngeal Movement Disorders in Multiple System Atrophy: A Diagnostic Biomarker? Mov Disord. 2020 Dec;35(12):2174-2183. doi: 10.1002/mds.28220. Epub 2020 Aug 5. PMID 32757231
- [Background] Gilman S, Wenning GK, Low PA, Brooks DJ, Mathias CJ, Trojanowski JQ, Wood NW, Colosimo C, Durr A, Fowler CJ, Kaufmann H, Klockgether T, Lees A, Poewe W, Quinn N, Revesz T, Robertson D, Sandroni P, Seppi K, Vidailhet M. Second consensus statement on the diagnosis of multiple system atrophy. Neurology. 2008 Aug 26;71(9):670-6. doi: 10.1212/01.wnl.0000324625.00404.15. PMID 18725592
- [Background] Hoglinger GU, Respondek G, Stamelou M, Kurz C, Josephs KA, Lang AE, Mollenhauer B, Muller U, Nilsson C, Whitwell JL, Arzberger T, Englund E, Gelpi E, Giese A, Irwin DJ, Meissner WG, Pantelyat A, Rajput A, van Swieten JC, Troakes C, Antonini A, Bhatia KP, Bordelon Y, Compta Y, Corvol JC, Colosimo C, Dickson DW, Dodel R, Ferguson L, Grossman M, Kassubek J, Krismer F, Levin J, Lorenzl S, Morris HR, Nestor P, Oertel WH, Poewe W, Rabinovici G, Rowe JB, Schellenberg GD, Seppi K, van Eimeren T, Wenning GK, Boxer AL, Golbe LI, Litvan I; Movement Disorder Society-endorsed PSP Study Group. Clinical diagnosis of progressive supranuclear palsy: The movement disorder society criteria. Mov Disord. 2017 Jun;32(6):853-864. doi: 10.1002/mds.26987. Epub 2017 May 3. PMID 28467028
- [Background] Isono C, Hirano M, Sakamoto H, Ueno S, Kusunoki S, Nakamura Y. Differential Progression of Dysphagia in Heredity and Sporadic Ataxias Involving Multiple Systems. Eur Neurol. 2015;74(5-6):237-42. doi: 10.1159/000442252. Epub 2015 Dec 1. PMID 26618669
- [Background] Kalf JG, de Swart BJ, Bloem BR, Munneke M. Prevalence of oropharyngeal dysphagia in Parkinson's disease: a meta-analysis. Parkinsonism Relat Disord. 2012 May;18(4):311-5. doi: 10.1016/j.parkreldis.2011.11.006. Epub 2011 Dec 3. PMID 22137459
- [Background] Laciuga H, Rosenbek JC, Davenport PW, Sapienza CM. Functional outcomes associated with expiratory muscle strength training: narrative review. J Rehabil Res Dev. 2014;51(4):535-46. doi: 10.1682/JRRD.2013.03.0076. PMID 25144167
- [Background] Mancopes R, Smaoui S, Steele CM. Effects of Expiratory Muscle Strength Training on Videofluoroscopic Measures of Swallowing: A Systematic Review. Am J Speech Lang Pathol. 2020 Feb 7;29(1):335-356. doi: 10.1044/2019_AJSLP-19-00107. Epub 2020 Jan 30. PMID 31999193
- [Background] Miller N, Noble E, Jones D, Burn D. Hard to swallow: dysphagia in Parkinson's disease. Age Ageing. 2006 Nov;35(6):614-8. doi: 10.1093/ageing/afl105. PMID 17047007
- [Background] Muller J, Wenning GK, Verny M, McKee A, Chaudhuri KR, Jellinger K, Poewe W, Litvan I. Progression of dysarthria and dysphagia in postmortem-confirmed parkinsonian disorders. Arch Neurol. 2001 Feb;58(2):259-64. doi: 10.1001/archneur.58.2.259. PMID 11176964
- [Background] O'Sullivan SS, Massey LA, Williams DR, Silveira-Moriyama L, Kempster PA, Holton JL, Revesz T, Lees AJ. Clinical outcomes of progressive supranuclear palsy and multiple system atrophy. Brain. 2008 May;131(Pt 5):1362-72. doi: 10.1093/brain/awn065. Epub 2008 Apr 2. PMID 18385183
- [Background] Panegyres PK, Hillman D, Dunne JW. Laryngeal dystonia causing upper airway obstruction in progressive supranuclear palsy. J Clin Neurosci. 2007 Apr;14(4):380-1. doi: 10.1016/j.jocn.2005.12.019. Epub 2006 Apr 4. PMID 16597502
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Silber MH, Levine S. Stridor and death in multiple system atrophy. Mov Disord. 2000 Jul;15(4):699-704. doi: 10.1002/1531-8257(200007)15:43.0.co;2-l. PMID 10928581
- [Background] Suttrup I, Warnecke T. Dysphagia in Parkinson's Disease. Dysphagia. 2016 Feb;31(1):24-32. doi: 10.1007/s00455-015-9671-9. Epub 2015 Nov 21. PMID 26590572
- [Background] Tilley E, McLoughlin J, Koblar SA, Doeltgen SH, Stern C, White S, Peters MD. Effectiveness of allied health therapy in the symptomatic management of progressive supranuclear palsy: a systematic review. JBI Database System Rev Implement Rep. 2016 Jun;14(6):148-95. doi: 10.11124/JBISRIR-2016-2002352. PMID 27532657
- [Background] Troche MS, Okun MS, Rosenbek JC, Musson N, Fernandez HH, Rodriguez R, Romrell J, Pitts T, Wheeler-Hegland KM, Sapienza CM. Aspiration and swallowing in Parkinson disease and rehabilitation with EMST: a randomized trial. Neurology. 2010 Nov 23;75(21):1912-9. doi: 10.1212/WNL.0b013e3181fef115. PMID 21098406
- [Background] Warnecke T, Suttrup I, Schroder JB, Osada N, Oelenberg S, Hamacher C, Suntrup S, Dziewas R. Levodopa responsiveness of dysphagia in advanced Parkinson's disease and reliability testing of the FEES-Levodopa-test. Parkinsonism Relat Disord. 2016 Jul;28:100-6. doi: 10.1016/j.parkreldis.2016.04.034. Epub 2016 Apr 28. PMID 27158122